CLINICAL TRIAL: NCT00279058
Title: The Role of Autologous Dendritic Cells Pulsed by Melanoma Associated Peptides to Augment the Therapeutic Effect of Interleukin-2
Brief Title: The Role of Peptide-loaded Dendritic Cells to Augment the Therapeutic Effect of Interleukin-2
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: pepDCIL2- HMO-CTIL
Record Dates: First submitted 2006-01-17; First posted 2006-01-19 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2007-04

CONDITIONS: Metastatic Melanoma
MeSH Terms: conditions — Melanoma

INTERVENTIONS:
Procedure: Immunotherapy treatment for melanoma

SUMMARY:
Melanoma is the main cause of death in patients with skin cancer. Once it has metastasized, this cancer has been shown to respond to chemotherapy only in rare cases. Immunotherapy represents an approach to treatment based on the immune response to cancer antigens.

The principal objective of the study is to identify whether a dendritic cell-based vaccine can increase the moderate therapeutic effect of bolus high dose IL-2 in patients with metastatic melanoma. For this purpose,patients with metastatic melanoma who have a certain blood type (HLA-A201+) will be treated systemically with high dose IL-2. In one group of patients, the IL-2 will be preceded by three doses of autologous dendritic cell pulsed with melanoma antigens appropriate for their blood type. Two cycles of three DC vaccines will be administered every 14 days by intra-lymph node injections, followed by high dose IL-2 treatment. Responding patients will receive additional DC vaccines at 1 month and 2 months intervals.

In a second group, patients will receive the standard high dose IL-2 protocol within a comparable period of time.

Each group will include 12 patients.

A complete evaluation of evaluable lesions will be performed prior to accrual, after initial 3 DC vaccines, six weeks after first IL-2 treatment, after a total of 6 DC vaccines and 6 weeks after second cycle of IL-2 treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Any patient age 18 to 65, with measurable metastatic melanoma who has an expected survival of greater than three months. All patients will be HLA-A2 positive

   * Patient must have received accepted standard treatmnet for melanoma - DTIC -containing protocol ,unless unwilling.
   * Patients who failed previous treatment with IL-2 will be included on a compassionate basis in the IL-2 plus vaccination scheme without being included in the analysis.
2. serum creatinine of 2.0 mg/dl or less,
3. Total bilirubin 1.6 mg/dl or less, except for patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dl.
4. WBC 3000/mm3 or greater
5. platelet count 90,000 mm3 or greater
6. serum AST/ALT less then two times normal
7. ECOG performance status of 0, 1 or 2.
8. Patients of both genders must be willing to practice effective birth control during this trial.
9. Patient agreed to participate in the study and has signed a written informed consent,
10. The patient must be eligible to receive IL-2.

Exclusion Criteria:

Patients will be excluded:

1. who are undergoing or have undergone in the past 3 weeks any other form of therapy except from surgery for their cancer.
2. have active systemic infections, coagulation disorders, autoimmune disease or other major medical illnesses of the cardiovascular or respiratory systems or any known immunodeficiency disease.
3. who require steroid therapy.
4. who are pregnant (because of possible side effects on the fetus).
5. who are known to be positive for hepatitis BsAG, HCV, or HIV antibody (because of possible immune effects of these conditions).
6. who have any form of primary or secondary immunodeficiency. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities.)
7. who are allergic to eggs.

i. who have an active major medical illnesses such as cardiac ischemia as evidenced by a stress thallium or comparable test, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease (to be eligible to receive IL-2 ) j. Have an abnormal thyroid function (to be eligible to receive IL-2).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2005-12; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Complete evaluation of untreated lesions with physical examination and appropriate X-rays and/or scans will be performed four to six weeks after the last DC injection.
Immunological evaluation will be performed two weeks after the last DC injection.

CONTACTS AND LOCATIONS:
Overall Officials: Michal Lotem, MD, Principal Investigator — Hadassah Medical Organization, pob 12000, Jerusalem, Israel
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel